CLINICAL TRIAL: NCT06578533
Title: Phase III, Multicenter, Open-label, Randomized Clinical Trial to Evaluate Efficacy of Sodium Zirconium Cyclosilicate (Lokelma) Compared to Standard of Care to Manage Hyperkalemia in Patients With Chronic Kidney Disease (CKD)
Brief Title: Keeping RAASi Treatment With Optimal Potassium Control
Acronym: KEEP-ON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-ON
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: Phase III multicenter, randomized, open-label, parallel-group non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients assigned to this group will have their iSRAA and/or ARM treatment withdrawn or reduced, according to standard clinical practice.
- Experimental group (Experimental): Patients assigned to this group will be maintained on treatment with iSRAA and/or ARM and oral treatment with CSZ (Lokelma) will be added. A single dose of CSZ consists of one to three sachets (5 to 10 g of active ingredient per sachet) that the subject must suspend in 45 mL of water.
  Interventions: Drug: Sodium Zirconium Cyclosilicate

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate — The recommended starting dose of Lokelma is 10 g, administered three times a day.
  If, at any time during the study, sK is > 6.5 mEq/L, treatment for acute hyperkalemia will be started following common clinical practice and local protocols, and investigator will consider RAASi / MRA withdrawal, or downtitration. In this case (confirmed sK > 6.5 mEq/L despite the maximum SZC dose) patient will leave the IP and will be counted as a treatment failure.
  If sK is ≤ 3.0 mEq/L, discontinue SZC. The subject should immediately receive appropriate medical intervention.
  If sK is between 3.1-5.1 mEq/L, pause SZC and re-evaluate in a week. This one-week SCZ treatment temporary discontinuation can only be applied once; if a new sK value between 3.1-5.1 mEq/L is detected, patient will leave the IP permanently.
  Depending on the serum potassium levels at each visit, the dose of SZC will be adjusted.
  Other Names: Lokelma
  Arms: Experimental group

SUMMARY:
Phase III, multicenter, randomized, open-label, parallel-group, non-inferiority, phase III clinical trial comparing CSZ (Lokelma) vs. iSRAA discontinuation/reduction and/or ARM (standard treatment).

DETAILED DESCRIPTION:
Hyperkalemia is a potentially life-threatening condition associated with ventricular arrhythmias and sudden cardiac arrest. It is common in patients with some comorbidities such as chronic kidney disease, congestive heart failure, cardiovascular disease, diabetes or liver disease. Most of these patients should receive drugs that block the renin angiotensin aldosterone system (RAASi) and mineralocorticoid receptor antagonists (MRA), that increase the risk of hyperkalemia.

For these reasons, relatively few patients receive maximum doses of RAASi / MRA. The dose and its usage decline following an hyperkalemia episode. However, RAASi / MRA discontinuation because of hyperkalemia, represents an undesirable clinical scenario, loosing their potential cardiorenal and nephroprotective benefit. Patients on submaximum doses or who discontinued RAASi / MRA have worse outcomes than patients on maximum doses.

In this study 78 adult patients will be randomized to one of two treatment arms to analyze the proportion of patients achieving sK of < 5.5 mEq/L:

* Control group: they will have their treatment with iSRAA and/or ARM withdrawn or tapered, according to standard clinical practice.
* Experimental group: treatment with iSRAA and/or ARM will be maintained and oral treatment with CSZ (Lokelma) will be added.

The study will be conducted in 3 periods:

* Patient selection (Visit 0).
* Randomization (Visit 1).
* Follow up (Visits 2-7).

All the patients randomized and completing the treatment assigned will be participating in the study for an stimated period of 90 ± 13 d. The clinical trial will be finalized when the last 90-day follow-up of the last patient included is performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must present serum potassium levels of 5.5-6.5 mEq/L at patient selection visit (V0)
* Patients must present serum potassium levels of 5.0-6.5 mEq/L at randomization visit (V1).
* Provision of patient or legal representative informed consent prior to any study specific procedures.
* Individuals receiving background standard of care for HF and treated according to locally recognized guidelines. Specific treatment should include RAASi and/or MRA treatment at first consultation and at least should have been stable for ≥ 4 weeks at maximum tolerated doses.
* Patients with CKD not on dialysis (Stages 2-5: estimated glomerular filtration rate (eGFR) between 15-60 ml/min/1,73m2 or eGFR between 60-90 ml/min/ 1.73 m2 with albuminuria/creatinuria (> 30 mg/g) in the previous three months). The estimated GFR can be reported by the laboratory or calculated by the researcher with serum creatinine, age, and sex (CKD-EPI equation).
* 18 years at the time of signing ICF.
* Negative pregnancy test (urine or serum) for female subjects of childbearing potential.
* Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign ICF) and for 3 months after the last dose of SZC. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
* Previous enrollment or randomization in the present study.
* HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy or uncorrected primary valvular disease.
* Current acute decompensated HF, hospitalization due to decompensated HF, myocardial infarction, unstable angina, stroke or transient ischemic attack within 12 weeks prior to enrollment.
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting or valvular repair/replacement within 12 weeks prior to enrollment or planned to undergo any of these operations after randomization).
* Implantation of a Cardiac Resynchronization Therapy (CRT) device or Implantable Cardioverter Defibrillator (ICD) within 12 weeks prior to enrollment or intent to perform atrial fibrillation ablation or to implant a CRT or ICD device.
* Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or transplantation or implantation expected after randomization
* Oropharingeal dysfunction that precludes normal swallow.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Patients with amputated limbs or pacemaker devices will be excluded of bioimpedance analysis.
* Participation in another clinical study with an investigational product during the last 6 months.
* Patients with a known hypersensitivity to SZC or any of the excipients of the product.
* Treated with potassium binding resins such as sodium polystyrene sulfonate (SPS; e.g. Kayexalate®) or calcium polystyrene sulfonate (CPS; e.g. Resonium®) or the cation exchange polymer, patiromer sorbitex calcium (Veltassa®), within 7 days prior to the first dose of study drug.
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.
* Subjects with a family history of long QT syndrome, presence of cardiac arrhythmias or conduction defects that require immediate treatment, or a QTc (corrected QT interval) of ≥ 550 msec.
* History of QT prolongation associated with other medications that required discontinuation of that medications.
* Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving serum potassium < 5.5mEq/L at three or all timepoints (7, 30, 60 or 90 days) after follow up (90 days) in both groups. | Through study completion, an average of 1 year
  To analyze the proportion of patients achieving sK of < 5.5 mEq/L with Sodium zirconium cyclosilicate (SZC) versus discontinuation of RAASi and/or MRA in patients with hyperkalemia and non dialysis CKD.

SECONDARY OUTCOMES:
Percentage of patients achieving serum potassium < 5 mEq/L at two of the four temporal points in both groups. | Through study completion, an average of 1 year
  To determine if the percentage of patients achieving serum potassium < 5 mEq/L at two of the four temporal points is not inferior in SZC compared to RAASi / MRA discontinuation or downtitration.
Number of patients treated with SZC with reduction of serum potassium > 20% after baseline in each time point. | Through study completion, an average of 1 year
  To determine the number of patients treated with SZC who effectively reduce serum potassium > 20 % over the baseline at days 7, 30, 60 and 90 compared to RAASi / MRA discontinuation or downtitration.
Percentage of patients achieving serum potassium below 5, 5.5, 6, 6.5 mEq/L in each time point. | Through study completion, an average of 1 year
  To compare percentage of patients achieving serum potassium below 5, 5.5, 6, 6.5 mEq/L at days 7, 30, 60 and 90 in both groups.
Percentage of patients requiring additional treatments for hyperkalemia in both groups (potassium binding resins, adding or increasing loop diuretics, or discontinuation of RAASi and/or MRA in Lokelma group. | Through study completion, an average of 1 year
  To compare the need for additional treatments for serum hyperkalemia between both groups during the study (potassium binding resins, adding or increasing loop diuretics if hypervolemia).
Mean change in the urine albumin-to-creatinine ratio (UACR) at 90 days from baseline in patients treated with SZC compared to RAASi / MRA discontinuation or downtitration. | Through study completion, an average of 1 year
  To compare albuminuria changes at 90 days from baseline.

OTHER OUTCOMES:
Mean and standard deviation comparation scores between groups at baseline and at the end of the study (visit 1 and 7) (MLHFQ and SF-36) | Through study completion, an average of 1 year
  To demonstrate an improvement in health-related quality of life in this patient population in patients treated with SZC when compared to the patients non treated with the drug.
Proportion of patients in each group with downtitration (decrease 25 %, 50 % 75 % or discontinuation of RAASi or MRI) during the study. | Through study completion, an average of 1 year
  To determine the number of patients treated with SZC who effectively need RAASi / MRA discontinuation or downtitration.
Difference between mean hydration percentage with respect to baseline (OH/ECV *100) measured by multifrequency bioimpedance (BCM, Fresenius) at 90 days. | Through study completion, an average of 1 year
  Changes in relative overhydration: (OH/ECV *100).
Proportion of patients treated with SZC presenting adverse events, in comparison to the patients non-treated with SZC, at 7, 30, 60 and 90 days | Through study completion, an average of 1 year
  To evaluate the safety and tolerability of SZC in relation to the patients non treated with the drug.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia

IPD SHARING:
Plan to Share IPD: Undecided